CLINICAL TRIAL: NCT06675565
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of ALN-AGT01 RVR in Adult Healthy Volunteers
Brief Title: A Study to Evaluate ALN-AGT01 RVR in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-AGT01 RVR-001
Record Dates: First submitted 2024-10-29; First posted 2024-11-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: RNAi therapeutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALN-AGT01 RVR (Experimental): Participants will be administered a single dose of ALN-AGT01 RVR.
  Interventions: Drug: ALN-AGT01 RVR
- Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-AGT01 RVR — ALN-AGT01 RVR will be administered subcutaneously (SC)
  Arms: ALN-AGT01 RVR
Drug: Placebo — Placebo will be administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and PK of single ascending doses of ALN-AGT01 RVR.

ELIGIBILITY:
Inclusion Criteria

* Is an adult healthy volunteer
* Has a body mass index ≥18 kg/m^2 and ≤28 kg/m^2

Exclusion Criteria

* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN)
* Has known human immunodeficiency virus infection; or known current or chronic hepatitis C virus or hepatitis B virus infection
* Has an estimated glomerular filtration rate (eGFR) of <90 mL/min/1.73m^2 at screening

Note: other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Up to 3 months

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of ALN-AGT01 RVR in Plasma | Predose and up to 3 days postdose
Maximum Observed Plasma Concentration (Cmax) of ALN-AGT01 RVR in Plasma | Predose and up to 3 days postdose
Time to Maximum Plasma Concentration (Tmax) of ALN-AGT01 RVR in Plasma | Predose and up to 3 days postdose
Concentrations of ALN-AGT01 RVR in Urine | Predose and up to 1 day postdone
  Fraction of ALN-AGT01 RVR excreted in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No